CLINICAL TRIAL: NCT01516034
Title: The Efficacy of the Cupola Ultrasonic Tattoo Removal Device: A Prospective Single Blinded, Before-After Study Design
Brief Title: The Efficacy of the Cupola Ultrasonic Tattoo Removal Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided that the results were not significant enough to continue.
Sponsor: Cupola Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR-2
Record Dates: First submitted 2012-01-16; First posted 2012-01-24 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-11

CONDITIONS: Tattooing
Keywords: Tattoo removal; ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Cupola Tattoo Removal Device
  Interventions: Device: Cupola Tattoo Removal device

INTERVENTIONS:
Device: Cupola Tattoo Removal device — Up to 6 treatments with the device every 2-3 weeks to the tattoo area.

SUMMARY:
The study is designed to determine the efficacy of the Cupola tattoo removal device for tattoo removal.

DETAILED DESCRIPTION:
The Cupola system is a non-invasive device for pigment/tattoo removal based on ultrasound technology. The safety of the device was demonstrated in a previous pilot study approved by the Herzog Helsinki committee #167-09, Ministry of Health April 2010 #HT-5293) showing that no risk was associated with the procedure.

This study is designed to determine the efficacy of the device for tattoo removal in up to 6 treatments in different treatment intervals. Three areas of the tattoo that are similar in size, color, and intensity will be chosen. One area will not be treated; the second will receive 6 treatments in 2-3 week intervals; the third will receive 3 treatments in 4-6 week intervals. The evaluations will include color measurements, photography, subject comfort and skin condition.

ELIGIBILITY:
Inclusion Criteria:

1. Tattoos

   * Age of tattoo - more than 1 year since application
   * Type - decorative (not cosmetic)
   * Not previously treated
2. General

   * At least 18 years of age
   * Agrees to sign the Informed Consent
   * Willingness to remove tattoo
   * Willingness to have photographs and color measurements of the treated area taken and to be used for marketing and educational presentation and/or publications
   * Willingness to follow the treatment schedule and post treatment care requirement for tattooing and removal
   * Not planning to remove the tattoo in a different procedure during the time of the experiment

Exclusion Criteria:

1. Skin conditions

   * Skin type 5 and 6
   * History of keloid formation
   * Active herpes simplex
   * Psoriasis or vitiligo
2. Other medical conditions

   * HIV or Hepatitis
   * Pregnancy or intention to become pregnant in the next 6 months
   * No allergic reaction during the tattooing process.
3. Medication

   * Currently taking anticoagulant medication, blood thinners, steroids or immunosuppressive
   * Taking isotretinoin (Accutane) currently or within the last 6 months
   * Minocyclin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Friedman, M.D., Principal Investigator — Friedman Skin & Laser Center; Lilach Gavish, Ph.D., Study Director — Friedman Skin & Laser Center
Locations (1):
- Dr David Friedman Laser & Skin Center, Diskin 60 st., Jerusalem, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 20-Nov-2011 to 11-Mar-12 Location: Dermatological clinic
Groups:
- Treatment: Cupola tattoo removal treatment
Period: Overall Study
Arm/Group | Treatment
Started | 8
Completed | 0
Not Completed | 8
Not completed — Physician Decision | 1
Not completed — Lack of Efficacy | 7

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.1 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  Israel | 8

OUTCOME MEASURES:

1. Primary Outcome: Tattoo Removal Efficiency
Description: Extent of Tattoo removal is quantified in 2 methods based on photographs taken at the baseline visit and at the termination visit:
  1. Scoring by independent dermatologist
  2. Measuring pigment clearance using image analysis
Time Frame: 6 months (termination)
Population: The number of participants that completed follow up.
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Tolerability Score
Description: The tolerability of the procedure will be scored by the subject using a Pain Visual Analog Scale on a 0 to 10 scale where 10 represents the highest degree of pain and 0 represents a complete lack of pain.
Time Frame: 0, 2, 4, 6, 8, 10 weeks (after every treatment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8)
Mild thickening of the skin (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days